CLINICAL TRIAL: NCT06255158
Title: The Effectiveness of an Individualized Intervention for Perpetrators of Child Sexual Abuse
Brief Title: Pilot Randomized Controlled Trial of the INSIGHT Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Marta Sousa, Principal Investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UID/01662/2020; 2020.06634.BD (Other Grant/Funding Number: Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2024-01-16; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Deviant Sexual Behavior
Keywords: effectiveness; RCT; child sexual abuse; schema therapy
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INSIGHT Program (Experimental): The design of the INSIGHT Program aligns with RNR model, the principles of cognitive behavioral therapy, and schema therapy. The intervention comprises different phases, beginning with an initial individual motivation interview intervention, and followed by a CBT-structured, ST-inspired individual program.
  The core of the intervention program consists of a manualized individual program comprising 25 weekly sessions, each lasting approximately 60 minutes.
  Interventions: Behavioral: INSIGHT Program
- Treatment As Usual Group (Other): TAU in Portuguese prisons is primarily aimed to increase educational and professional qualifications
  Interventions: Other: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: INSIGHT Program — INSIGHT Program:
  the program targets the reduction of EMSs' interference in social information processing, which may otherwise lead to the use of deviant behavior to fulfill emotional and sexual needs. Furthermore, the program has specific goals: (1) developing insight about the offense cycle; (2) fostering empathy for victims; (3) enhancing intimate and social/ interpersonal skills; (4) increasing emotional regulation skills.
  Arms: INSIGHT Program
Other: Treatment As Usual (TAU) — TAU in Portuguese prisons is primarily aimed to increase educational and professional qualifications
  Arms: Treatment As Usual Group

SUMMARY:
This randomized controlled trial aimed to assess the efficacy of a new intervention program for perpetrators of child sexual abuse: the INSIGHT Program. The primary outcome measures to assessing INSIGHT effectiveness will include psychological symptoms, EMSs, cognitive distortions, interpersonal problems, self-esteem, victim empathy, and empathy, and sexual violence risk. Then, qualitative interviews will enable an in-depth examination of the therapeutic process and its effects.

DETAILED DESCRIPTION:
Perpetrators of CSA will be recruited from Portuguese Prisons. Potential participants who are likely to meet inclusion criteria will be identified and referred to study staff by prison members.

Participants who agreed to participate gave written informed consent, completed the baseline assessment, and were randomly assigned to treatment conditions (treatment and control groups) using a random number table by a research assistant who was blind to any information about each participant.

Besides baseline assessment, participants completed the post-treatment assessment (at the end of INSIGHT Program) and follow-up assessment (3 months after INSIGHT completion).

The program's structured and manualized design ensures integrity, at least partially.

ELIGIBILITY:
Inclusion Criteria:

* male;
* men with convictions of a sexual crime against a child

Exclusion Criteria:

* men with cognitive disabilities;
* men with psychotic symptoms;
* men with higher traits of psychopathy;
* men with addiction to alcohol/drugs;
* men with convictions for child pornography and/or rape (i.e., adult victims)
* men in prison less than 12 months since the beginning of the program
* Female;
* men having low risk of sexual recidivism

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Hanson Sex Attitude Questionnaire (HSAQ; Hanson et al., 1994; Portuguese version by Sousa et al., in press) | immediately post-intervention and 3-month follow-up
  The study protocol will include the Hanson Sex Attitude Questionnaire (HSAQ; Hanson et al., 1994; Portuguese version by Sousa et al., in press). The Portuguese version of HSAQ is a 38-items self-report measure designed to measure cognitive distortions about child sexual abuse and sexuality. Through a confirmatory factor analysis, it was possible to identify three independent factors, namely: Child as human beings (17 items), Sexual Drive (12 items), and Sexual entitlement (9 items). Each item is scored on a 5-point ordinal scale (1 = strongly disagree to 5 = strongly agree). The scale does not have a cutoff point, but higher scores indicated more cognitive distortions. In factor 1, scores can vary between 17 and 85, in factor 2 from 12 to 60 and in factor 3 from 9 to 45.
Victim Empathy Distortion Scale (VES; Beckett & Fisher, 1994; Portuguese version: Sousa et al., in press) | immediately post-intervention and 3-month follow-up
  The study protocol will include the Victim Empathy Distortion Scale (VES; Beckett & Fisher, 1994; Portuguese version: Sousa et al., in press. VES is a 28-item questionnaire to assess the individual's understanding of the impact of offending on their victims. The Portuguese version of the scale has two factors: positive misattributions of pleasure in sexual abuse (18 items), and negative attributions of child sexual abuse (10 items). The scale does not have a cutoff point but higher scores on factor one indicated more cognitive distortions about child sexual abuse, while a higher score in factor 2 represents a greater awareness of the impact that the abusive situation has on their victim. The items are rated on a 5-point scale ranging from 0 (strongly disagree) to 4 (strongly agree). In factor 1, scores can vary between 18 and 90, in factor 2 between 10 and 50.
Basic Empathy Scale - Adapted (BES Adapted; Salas-Wright et al., 2012; Portuguese version: Pechorro et al., 2015). | immediately post-intervention and 3-month follow-up
  The study protocol will include the Basic Empathy Scale - Adapted (BES Adapted; Salas-Wright et al., 2012; Portuguese version: Pechorro et al., 2015). The BES Adapted is a self-report measure with two dimensions: affective empathy which encompasses three items, and cognitive empathy which includes four items. Each item is scored on a 5-point ordinal scale (1 = strongly disagree to 5 = strongly agree). The scale does not have a cutoff point, but higher scores indicate greater empathy. In the "affective empathy" factor, scores can vary between 3 and 15, in the "cognitive empathy" factor between 4 and 20. The total score can vary between 7 and 35.
Rosenberg Self-Esteem Scale (RSES; Rosenberg, 1979, 1989; Portuguese version: Pechorro et al., 2011). | immediately post-intervention and 3-month follow-up
  The study protocol will included the Rosenberg Self-Esteem Scale (RSES; Rosenberg, 1979, 1989; Portuguese version: Pechorro et al., 2011). RSES is a brief self-report scale that assesses self-esteem. Responses are coded on a 4-point scale ranging from 0 (strongly disagree) to 3 (strongly agree). the scale does not have a cutoff point, but higher results reveal higher levels of self-esteem. The total score can vary between 0 and 30.
Inventory of Interpersonal Problems (IIP-32; Barkham et al., 1996; Portuguese version by Faustino & Vasco, 2020). | immediately post-intervention and 3-month follow-up
  IIP-32 is a self-report instrument that focuses on the assessment of eight interpersonal domains: domineering/controlling; intrusive-needy; self-sacrificing; overly accommodating; nonassertive; socially avoidant ; cold-distant; and vindictive/self-centered. It is composed by 32 items rated along a 5-point Likert type scale response. No normative data are available.
Young Schema Questionnaire - YSQ-S3 (Young, 2005; Portuguese version by Pinto-Gouveia, Rijo, & Salvador, unpublished). | immediately post-intervention and 3-month follow-up
  The study protocol will include the Young Schema Questionnaire - YSQ-S3 (Young, 2005; Portuguese version by Pinto-Gouveia, Rijo, & Salvador, unpublished). The YSQ-S3 is a self-report questionnaire comprising 90 items. It measures 18 different EMS proposed by Young (1990) using a 6-point type scale (1 = completely untrue to me; 6 = to describe me perfectly). We generally consider any score of 3 or more on a schema to be meaningful. The total score can vary between 0 and 6.
Brief Symptoms Inventory (BSI; Derogatis, 2001; Portuguese version: Canavarro, 2007). | immediately post-intervention and 3-month follow-up
  The study protocol will include the Brief Symptoms Inventory (BSI; Derogatis, 2001; Portuguese version: Canavarro, 2007). BSI is a 53-item self-report instrument that measures psychopathological symptoms during the previous 7 days, on a five-point scale (0 = not at all to 4 = extremely). The inventory was composed of nine dimensions: somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. The cut-off point for the somatization scale is 0.6, for the obsessions-compulsions scale is 1.6, for the interpersonal sensitivity scale is 1.1, for the depression scale is 1.2, for the anxiety scale is 1.3, for the hostility scale is 1.1, for the phobic anxiety scale is 0.6, for the paranoid ideation scale is 1.3, and for the psychoticism scale is 0.9 (Canavarro, 2007). The total score can vary between 0 and 4.
Sexual Violence Risk (SVR-20; Boer et al., 1997; Portuguese version: Gonçalves & Vieira, 2004). | immediately post-intervention and 3-month follow-up
  SVR-20 is a structured professional judgment assessment instrument intended for use with perpetrators of sexual crimes. The instrument contains 20 items that are considered risk factors for recidivism in sexual crimes. Professionals use clinical judgment and file information to rate each of the 20 items as either "not present", "possibly or partially present" or "present". The instrument contains three sections: psychosocial adjustment (7 items), sex offenses (7 items) and future plans (2 items). the scale does not have a cutoff point.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minho, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT06255158/SAP_000.pdf
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT06255158/ICF_001.pdf